CLINICAL TRIAL: NCT01146561
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH CHRONIC PANCREATITIS
Brief Title: Safety And Efficacy Of Tanezumab In Patients With Chronic Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091044; 2010-019012-21 (EudraCT Number); CHRONIC PANCREATITIS POC STUDY (Other: Alias Study Number)
Record Dates: First submitted 2010-05-24; First posted 2010-06-17 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tanezumab 20 mg (Experimental)
  Interventions: Biological: Tanezumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tanezumab — single administration of tanezumab 20 mg sub-cutaneously
  Arms: Tanezumab 20 mg
Other: Placebo — single administration of placebo to match tanezumab, sub-cutaneously
  Arms: Placebo

SUMMARY:
Tanezumab is effective in reducing the pain associated with chronic pancreatitis.

DETAILED DESCRIPTION:
On 23 Dec 2010 the FDA imposed a clinical halt for anti-NGF compounds due to safety reasons, ie, a case of osteonecrosis which occurred in relation to an anti-NGF compound of another company. All indications with the exception of Cancer Pain are affected resulting in termination of all studies in respective indications. Recruitment of Study A4091044 was stopped effective 27 Dec 2010. Two patients recruited so far did not receive further doses and were followed up for safety until LSLV on 22 Mar 2011.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Written informed consent
* Diagnosis of chronic pancreatitis based on imaging studies
* Persistent abdominal pain due to chronic pancreatitis
* Qualifying pain score during the pre-treatment period
* Willing to comply with study visit schedule and study requirements including for women of child-bearing potential or male patients with female partners of child-bearing potential, the use of 2 forms of birth control

Exclusion Criteria:

* Pregnant women, lactating mothers, women suspected of being pregnant and women who wish to become pregnant during the course of the study
* Chronic pancreatitis as a complication of pancreatic cancer or acute pancreatic duct obstruction
* Pancreatic surgery, lithotripsy or endoscopist decompression within 3 months
* History of alcoholism (within 1 year of screening) or concurrent alcohol abuse
* History of cancer in the past years
* Significant cardiac disease within 6 months
* History, diagnosis or signs and symptoms of significant neurologic disease
* Disqualifying laboratory values including Hepatitis B or C, HIV and drug test
* Other medical condition that may interfere with study endpoints or safety of the patient as determined by the Investigator
* Known history of rheumatoid arthritis
* Avascular necrosis of the bone
* History of trauma to a major joint Evidence of osteoarthritis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10-13 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2011-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Gastroenterology Group-of Naples, Naples, Florida
  - Palm Beach Gastroenterology, Wellington, Florida
  - Digestive Health Specialists, Tupelo, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Carolinas Digestive Health Associates, Harrisburg, North Carolina
  - UMPC Division of Radiology, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091044&StudyName=Safety%20And%20Efficacy%20Of%20Tanezumab%20In%20Patients%20With%20Chronic%20Pancreatitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the United States Food and Drug Administration (FDA) clinical hold, the study was prematurely terminated and no participants were enrolled in planned reporting arm tanezumab 20 milligram (mg) treatment and hence tanezumab 20 mg could not be administrated.
Groups:
- Placebo: A single dose of placebo matched to tanezumab 20 milligram (mg) injection subcutaneously on Day 1.
Period: Overall Study
Arm/Group | Placebo
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Placebo
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 1
  45 to 64 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Chronic Pancreatitis Pain Intensity Score Over the Period From Week 1 to Week 8
Description: Daily average chronic pancreatitis pain is assessed with an 11-point Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 1 to 8
Population: No efficacy analysis were performed as no tanezumab participant and only two placebo participants were randomized due to early study discontinuation of FDA clinical hold.
Arm/Group | Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Average and Worst Chronic Pancreatitis Pain Intensity Score at Week 1, 2, 4, 6, 8, 12 and 16
Description: Daily average chronic pancreatitis pain and worst chronic pancreatitis pain are assessed with an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Worst Chronic Pancreatitis Pain Intensity Score Over Week 1 to Week 8 Period
Description: Daily average worst chronic pancreatitis pain is assessed with an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 1 to 8
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With At Least 30 Percent (%), 50%, 70% and 90% Reduction From Baseline in Average and Worst Chronic Pancreatitis Pain Intensity Score
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Average and Chronic Pancreatitis Pain Intensity Score
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory - Short Form (BPI-sf) Average and Worst Pain Score at Week 8 and 16
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf are 4 questions that assess pain intensity (question 5 consists of 7 items that assess level of interference of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure were scored by item, with lower scores indicated less pain or pain interference.
Time Frame: Baseline, Week 8, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory - Short Form (BPI-sf) Pain Interference Index and Pain Interference Score for General Activity, Walking Ability, Sleep and Normal Work at Week 8 and 16
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf are 4 questions that assess pain intensity (worst, least, average, right now) and question 5 consisted of 7 items that assess level of interference of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure was scored by item, with lower score indicated less pain or pain interference. The 7 items in question 5 were averaged to obtain pain interference index, range: 0 to 10; higher score=greater impairment.
Time Frame: Baseline, Week 8, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Chronic Pancreatitis at Week 4, 8 and 16
Description: Patient's Global Assessment of Chronic Pancreatitis is a global evaluation that utilizes a 5-point Likert scale with a score of 1 being the best (Very Good) and a score of 5 being the worst (Very Poor) for the following question: "Considering all the ways your chronic pancreatitis affects you, how are you doing today?".
Time Frame: Baseline, Week 4, 8, 12
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Improvement of Greater Than or Equal to 2 Points From Baseline in Patient's Global Assessment (PGA) of Chronic Pancreatitis
Description: as for outcome 8
Time Frame: Weeks 4, 8, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Anti Drug Antibody
Time Frame: Baseline, Week 8, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

11. Secondary Outcome: Neuropathy Impairment Score (NIS)
Description: NIS: 74-item questionnaire assesses muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS score range 0-244, higher score=greater impairment.
Time Frame: Baseline and Weeks 2, 4, 8, 16
Population: as for outcome 1
Arm/Group | Placebo
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Injection Site Reaction
Description: Assessment of the injection site reactions were based on presence of erythema (redness), induration (swelling), ecchymosis (bruising), pruritus (itching) and pain that occurred after the injection had been administered (not related to pain of needle insertion).
Time Frame: Day 1 up to Week 16
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 2
Participants | 1

13. Secondary Outcome: Plasma Tanezumab Levels
Time Frame: Baseline (pre-dose), Week 2, 4, 8, 16
Population: No pharmacokinetic analysis were performed as no tanezumab participant and only two placebo participants were randomized due to early study discontinuation of FDA clinical hold.
Arm/Group | Placebo
Number analyzed (Participants) | 0

14. Secondary Outcome: Serum Nerve Growth Factor (NGF) Levels
Time Frame: Baseline (pre-dose), Week 8, 16
Population: No analysis was performed for this outcome measure as no tanezumab participant and only two placebo participants were randomized due to early study discontinuation of FDA clinical hold.
Arm/Group | Placebo
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 112 days after the dose of study medication (up to 113 days)
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 2
Participants
  AEs | 2
  SAEs | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory analysis included blood chemistry, hematology, urinalysis, pregnancy test, glycosylated hemoglobin levels (HbA1c levels) test and blood alcohol test.
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 2
Participants | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: All standard intervals (PR, QRS, QT, QT interval corrected for heart rate using Fridericia's formula [QTcF], QT interval corrected for heart rate using Bazett's formula [QTcB], RR intervals and heart rate) were analyzed for ECG abnormalities.
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 2
Participants | 0

18. Other Pre Specified Outcome: Number of Participants With Subcutaneous Doses
Description: Number of participants who received the single dose of placebo are reported.
Time Frame: Day 1
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2)
Injection site reaction (General disorders) | 1
Pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Due to FDA clinical hold, the study was prematurely terminated with only 2 participants were enrolled and randomized to placebo treatment and hence, efficacy and pharmacokinetic analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.